CLINICAL TRIAL: NCT00072020
Title: Does Adjuvant Zoledronic Acid Reduce Recurrence in Patients With High Risk Localized Breast Cancer?
Brief Title: Chemotherapy and/or Hormone Therapy With or Without Zoledronate in Treating Women With Stage II or Stage III Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sheffield (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: SHEFF-AZURE; CDR0000335111 (Registry Identifier: PDQ (Physician Data Query)); EU-20315; ISRCTN79831382; BIG-1-04
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2006-01

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: bone metastases; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Zoledronic Acid; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: zoledronic acid
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Zoledronate may delay or prevent the formation of bone metastases. It is not yet known whether chemotherapy and/or hormone therapy are more effective with or without zoledronate in preventing cancer recurrence and bone metastases in women with breast cancer.

PURPOSE: This randomized phase III trial is studying giving chemotherapy and/or hormone therapy together with zoledronate to see how well they work compared to chemotherapy and/or hormone therapy alone in preventing cancer recurrence and bone metastases in women with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare disease-free survival of women with stage II or III breast cancer at high risk of relapse treated with neoadjuvant or adjuvant chemotherapy and/or hormonal therapy with vs without zoledronate.

Secondary

* Compare time to bone metastases, as first recurrence, in patients treated with these regimens.
* Compare time to bone metastases, per se, in patients treated with these regimens.
* Compare time to distant metastases in patients treated with these regimens.
* Compare overall survival in patients treated with these regimens.
* Compare the reduction in skeletal-related events (fractures, spinal cord compression, radiotherapy to the bone, surgery to the bone, and hypercalcemia) before and after the development of bone metastases in patients treated with these regimens.
* Determine the safety and toxicity of zoledronate in patients treated with these regimens.
* Correlate prognostic factors, such as estrogen-receptor and progesterone-receptor status, TNM stage, tumor grade, HER2/neu status, and menopausal status with treatment outcome in patients treated with these regimens.
* Determine more specific prognostic indicators for the development of bone metastases and factors that are able to predict specific benefit from bisphosphonate treatment using proteomics, tissue micro-array, and other modern techniques in these patients.

OUTLINE: This is a randomized, open-label, parallel-group, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive neoadjuvant or adjuvant chemotherapy and/or hormonal therapy. Patients also receive concurrent zoledronate IV over 15 minutes every 3-4 weeks for 6 doses, every 3 months for 8 doses, and then every 6 months for 5 doses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive neoadjuvant or adjuvant chemotherapy and/or hormonal therapy alone.

After completion of study treatment, patients are followed annually for 5 years.

PROJECTED ACCRUAL: A total of 3,300 patients (1,650 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary breast cancer, meeting 1 of the following staging criteria:

  * Stage II
  * Stage III
  * T stage ≥ T1
* Receiving OR scheduled to receive chemotherapy and/or endocrine therapy

  * For patients receiving neoadjuvant therapy

    * Tumor > 5 cm (T3), features of locally advanced disease (T4), OR biopsy-proven lymph node involvement (N1)
    * Scheduled to proceed to definitive surgery and/or radical radiotherapy with curative intent within 6 months of starting neoadjuvant therapy
    * No more than 30 days between initiation of neoadjuvant therapy and start of study drug
  * For patients receiving adjuvant therapy

    * Must have undergone complete primary tumor resection and treatment of axillary lymph nodes*
    * Must have lymph node involvement
    * No prior neoadjuvant therapy**
    * No more than 60 days since prior definitive surgery NOTE: *Patients whose treatment plan includes further primary tumor resection and/or treatment of the axillary lymph nodes (e.g., clearance or radiotherapy) with curative intent after completion of chemotherapy are eligible provided the treatment is completed within 9 months of study entry

NOTE: **Preoperative endocrine therapy with a duration of < 30 days is not considered prior neoadjuvant therapy

* No evidence of recurrent or metastatic disease
* No history of breast cancer, except ductal carcinoma in situ or lobular carcinoma in situ
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Premenopausal or postmenopausal

Performance status

* Karnofsky 80-100% OR
* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Creatinine ≤ 1.5 times upper limit of normal

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active dental problems, including dental abscess or infection of the jaw bone (e.g., maxilla or mandible)
* No prior or current diagnosis of osteonecrosis of the jaw
* No other malignancy within the past 5 years (including prior contralateral breast cancer) except nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No history of disease with influence on bone metabolism, including any of the following:

  * Paget's disease of the bone
  * Primary hyperparathyroidism
  * Osteoporosis requiring treatment or likely to require treatment within the next 6 months
* No other severe physical or psychological disease that would preclude study compliance
* No known hypersensitivity to bisphosphonates

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* More than 4 weeks since prior and no concurrent dental or jaw surgery (e.g., extractions or implants)

  * Dental fillings, teeth scaling and polishing, or minor gingival surgery within the past 4 weeks are allowed

Other

* More than 1 year since prior bisphosphonates
* More than 30 days since prior investigational drugs
* No concurrent investigational drugs (i.e., not locally approved for any indication)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08

PRIMARY OUTCOMES:
Disease-free survival as assessed annually for 10 years

SECONDARY OUTCOMES:
Time to bone metastases as first recurrence assessed annually for 10 years
Time to bone metastases per se as assessed annually for 10 years
Time to distant metastases as assessed annually for 10 years
Overall survival as assessed by final analysis at 10 years
Skeletal-related events prior to development of bone metastases as assessed annually for 10 years
Skeletal-related events following development of bone metastases as assessed annually for 10 years
Safety and toxicity of zoledronic acid as assessed annually for 10 years
Evaluation of the influence of prognostic factors (e.g., estrogen receptor or progesterone receptor [ER/PR] status, TNM stage, tumor grade, HER2/neu, and menopausal status) on treatment outcome
Analysis of tumor-specific mutations, proteomics and gene expression changes in tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Coleman, MD, FRCP — Cancer Research Centre at Weston Park Hospital; Victoria Hiley — University of Leeds

REFERENCES:
- [Result] Marshall H, Gregory W, Bell R, et al.: Adjuvant therapy with zoledronic acid (AZURE-BIG 01/04): The influence of menopausal status and age on treatment effects. [Abstract] J Clin Oncol 30 (Suppl 15): A-502, 2012.
- [Result] Coleman RE, Marshall H, Cameron D, Dodwell D, Burkinshaw R, Keane M, Gil M, Houston SJ, Grieve RJ, Barrett-Lee PJ, Ritchie D, Pugh J, Gaunt C, Rea U, Peterson J, Davies C, Hiley V, Gregory W, Bell R; AZURE Investigators. Breast-cancer adjuvant therapy with zoledronic acid. N Engl J Med. 2011 Oct 13;365(15):1396-405. doi: 10.1056/NEJMoa1105195. Epub 2011 Sep 25. PMID 21995387
- [Result] Coleman R, Woodward E, Brown J, Cameron D, Bell R, Dodwell D, Keane M, Gil M, Davies C, Burkinshaw R, Houston SJ, Grieve RJ, Barrett-Lee PJ, Thorpe H. Safety of zoledronic acid and incidence of osteonecrosis of the jaw (ONJ) during adjuvant therapy in a randomised phase III trial (AZURE: BIG 01-04) for women with stage II/III breast cancer. Breast Cancer Res Treat. 2011 Jun;127(2):429-38. doi: 10.1007/s10549-011-1429-y. Epub 2011 Mar 11. PMID 21394500
- [Result] Coleman RE, Winter MC, Cameron D, Bell R, Dodwell D, Keane MM, Gil M, Ritchie D, Passos-Coelho JL, Wheatley D, Burkinshaw R, Marshall SJ, Thorpe H; AZURE (BIG01/04) Investigators. The effects of adding zoledronic acid to neoadjuvant chemotherapy on tumour response: exploratory evidence for direct anti-tumour activity in breast cancer. Br J Cancer. 2010 Mar 30;102(7):1099-105. doi: 10.1038/sj.bjc.6605604. Epub 2010 Mar 16. PMID 20234364
- [Result] Coleman R, Thorpe H, Cameron D, et al.: Zoledronic acid is well tolerated and can be safely administered with adjuvant chemotherapy first safety data from the AZURE trial (BIG01/04). [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-2080, S107, 2006.
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Coleman R, Cameron D, Dodwell D, Bell R, Wilson C, Rathbone E, Keane M, Gil M, Burkinshaw R, Grieve R, Barrett-Lee P, Ritchie D, Liversedge V, Hinsley S, Marshall H; AZURE investigators. Adjuvant zoledronic acid in patients with early breast cancer: final efficacy analysis of the AZURE (BIG 01/04) randomised open-label phase 3 trial. Lancet Oncol. 2014 Aug;15(9):997-1006. doi: 10.1016/S1470-2045(14)70302-X. Epub 2014 Jul 15. PMID 25035292